CLINICAL TRIAL: NCT06374563
Title: Tackling Chronic Pressure Ulcer Via Bee Venom Phonophoresis
Brief Title: Tackling Pressure Ulcer Via Bee Venom Phonophoresis
Acronym: ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Reham Alaa, lecturer of physical therapy, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BUC-IACUC-221109-6
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Bee Venom; Pressure Ulcers; Phonophoresis
Keywords: phonophoresis; bee venom
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Group 1 received topical application of Bee Venom gel, 3 times per week
  Interventions: Other: group 1 received topical Bee venom gel
- group 2 (Experimental): Group 1 received phonophoresis of Bee Venom gel using low intensity ultrasound, 3 times per week
  Interventions: Other: Group 2: Phonophoresis of Bee Venom gel

INTERVENTIONS:
Other: group 1 received topical Bee venom gel — Group 1 received a topical application of Bee Venom gel, 3 times per weeks. The wound dressing changed day after day and was cleaned every time with normal saline.
  Arms: Group 1
Other: Group 2: Phonophoresis of Bee Venom gel — group 2 received phonophoresis of Bee Venom gel using low frequency ultrasound, 3 times per weeks
  Arms: group 2

SUMMARY:
This study aimed to investigate the efficiency of topical Bee Venom gel versus phonophoresis of Bee Venom gel to accelerate healing of chronic pressure ulcer

DETAILED DESCRIPTION:
In this study, the Bee Venom gel was prepared in a gel formula. Patients with chronic pressure ulcers were enrolled randomly into two different groups. Group 1 received a topical application of Bee Venom gel, 3 times per weeks. While group 2 received phonophoresis of Bee Venom gel using low frequency ultrasound, 3 times per week. The treatment lasted for 8 consecutive weeks. The Image J Software is used to measure the wound surface area before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patients with stage II and III chronic neuropathic ulcers.

Exclusion Criteria:

* Patients with chronic cardiac,
* Patients with renal, and
* Patients with hepatic diseases and
* Diabetic patients. Additionally,
* Patients with immunosuppressive diseases,
* Patients with HIV, and
* Anemia Patients

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
wound surface area wound surface area | Before starting treatment and after 8 weeks of treatment
  ImageJ Software was used to measure the wound size
wound volume | Before starting treatment and after 8 weeks of treatment
  wound volume was measured through the volumetric measurement method using a syringe filled with saline

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Hassan, professor, Study Director — Badr University in Cairo
Locations (1):
- Badr University in Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No